CLINICAL TRIAL: NCT03575117
Title: Views on Colorectal Cancer Beliefs, Colorectal Cancer Worry, and Physical Activity
Brief Title: Views on Cancer Prevention and Daily Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Responsible Party: Principal Investigator, Linda Diane Cameron, Professor and Chair of Psychological Sciences, University of California, Merced
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCM2018-1
Record Dates: First submitted 2018-03-15; First posted 2018-07-02 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Sedentary Lifestyle
MeSH Terms: conditions — Colorectal Neoplasms; Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCI HYT--GA + CSM--Be Well (Experimental): Participants who view the Common Sense Model (CSM) "Be Well" text and image communication will be invited to receive two sets of daily text messages: (1) one text message and one image per day and (2) National Cancer Institute (NCI) HealthyYouTXT-Get Active (HYT-GA) program that is delivered 2-5 times daily for 6 weeks. After baseline and at timepoint 2, participants will view a slide presentation with imagery and text related to colorectal cancer risk and sedentary lifestyle. The same messages will be delivered as a drip campaign alongside the NCI HYT-GA text messaging program.
  Interventions: Behavioral: Common-Sense Model (CSM) Be Well; Behavioral: NCI HealthyYouTXT--Get Active (HYT--GA)
- NCI HYT--GA + ACS usual messages (Other): Adapted American Cancer Society (ACS) informational messages about colorectal cancer risk and lifestyle will be invited to receive one set of daily text messages, NCI HealthyYouTXT-Get Active (HYT-GA) program that is delivered 2-5 times daily for 6 weeks. After baseline and at timepoint 2, participants will view an informational slide presentation that is based on adapted language from American Cancer Guidelines related to cancer prevention and physical activity (https://www.cancer.org/healthy/eat-healthy-get-active/acs-guidelines-nutrition-physical-activity-cancer-prevention.html).
  Interventions: Behavioral: ACS usual messages; Behavioral: NCI HealthyYouTXT--Get Active (HYT--GA)

INTERVENTIONS:
Behavioral: Common-Sense Model (CSM) Be Well — Theoretically informed text messages and images that cover how physical activity is linked to decreasing colorectal cancer risk.
  Arms: NCI HYT--GA + CSM--Be Well
Behavioral: ACS usual messages — Information distributed by the American Cancer Society as information on the link between physical activity and cancer risk (source: www.cancer.org)
  Arms: NCI HYT--GA + ACS usual messages
Behavioral: NCI HealthyYouTXT--Get Active (HYT--GA) — Text messaging program developed by National Cancer Society (NCI). It is a free SMS program that promotes physical activity.

SUMMARY:
This study is to assess how a theoretically guided mHealth communication informed by evidence of thoughts and affect about colorectal cancer can enhance how an existing mHealth (cell/mobile based text messaging health promotion) intervention increased physical activity in healthy adults.

DETAILED DESCRIPTION:
Guided by the Common-Sense Model (CSM) of self-regulation and informed by prior evidence or knowledge about cancer beliefs and response to cancer risk, the investigators have now developed a complementary text and imagery based health communication called CSM--Be Well. During 2017, researchers completed three waves of data collection and pilot research that included: (a) cognitive interviews during Spring 2017, (b) manipulation check of initial health communication during Summer 2017, and (c) manipulation and quality check of final draft of health communication during Fall 2017. In this process and guided by the CSM, the investigators have developed a library of text and images (CSM--Be Well) based on information that increases understanding of colorectal cancer risk and promotes physical activity as a protective behavior against colorectal cancer. CSM--Be Well has been created as 36-slide presentation. In addition, each slide serves as a daily text message.

The purpose of the present research is to evaluate the appropriateness of our final CSM--Be Well health communication and how it enhances the National Cancer Society's HealthyYouTXT--Get Active (HYT--GA) program. To examine how well it increases understanding colorectal cancer risk and promotes physical activity, it will be compared to usual care information based on the American Cancer Society's (ACS) usual messages promoting cancer prevention and protective behaviors (i.e., physical activity, diet, and alcohol intake).

The research design is a 6-week, longitudinal, randomized control trial with two arms: experimental and control. All participants are asked to sign up for HYT--GA 6-week text messaging program. The experimental arm will view the CSM--Be Well program as a slide presentation on a website. Also, they will receive a daily drip campaign of the parsed slides that were seen at baseline activities. The control arm will view the ACS usual text as a slide presentation on a website.

In addition, the investigators will conduct surveys to evaluate the appropriateness of the theoretical framework on which the CSM--Be Well program is based. Participants will be asked to complete surveys at 8 timepoints. At enrollment (Baseline; Timepoint 1), participants will be invited to view, 2 to 3 days later (Timepoint 2), an informational session on colorectal cancer prevention and physical activity (CSM--Be Well or ACS usual messages) and to sign-up for a 6-weeks daily text messages (HYT--GA). In addition, researcher will conduct surveys to evaluate responses and user engagement. After 1 week (Timepoint 3), participants will be invited to complete surveys with measures of their understanding of colorectal cancer risk, measures of coherent understanding of colorectal cancer, physical activity behavior in the past week and future plans, and risks, concerns, and worries about colorectal cancer risk. These survey responses will be used to compare how values and self-regulation factors distinctively predict physical activity motivations and behaviors. After 2 weeks (Timepoints 3 to7), participants will be asked 5 times to a weekly brief surveys about their past and future physical activity levels. After 6 weeks (Timepoint 8), participants will be invited to complete final survey with measures of their understanding of colorectal cancer risk, measures of coherent understanding of colorectal cancer, physical activity behavior in the past week and future plans, and risks, concerns, and worries about colorectal cancer risk.

ELIGIBILITY:
Inclusion Criteria:

1. Open to all interested who are 18 years of age and older, all genders, all ethnic and/or racial identities, and regardless of health status.
2. Capacity to engage in physical active without medical and/or assisted supervision. During screening, this will be assessed by the Physical Activity Readiness (PAR-Q) survey. It confirms capacity to engage in physical activity that does not need to be medically/professionally supervised.
3. Has interest and ability to receive Short Message Service (SMS) text messages linked to a cell phone and access to the internet for information that is web based.
4. Individuals who report light/moderate physically active and sedentary lifestyles (<6.0 METs). METs are the metabolic equivalents that measures the energy related to physical activity and/or sedentary behavior.
5. Interest in wearing a pedometer.

Exclusion Criteria:

1. Reports of vigorous levels of physical activity. Specifically, those who report >6.0 METs. METs are the metabolic equivalents that measures the energy related to physical activity and/or sedentary behavior.
2. Those who report that a medical doctor has recommended anytime with the last 12 months that there be limited physical activity due to heart disease, pain, physical ailments, dizziness, loss of consciousness, bone/joint problems related to engaging in physical activity.
3. Those who report that a doctor recommended against engaging in supervised physical activity and/or moderate physical activity (such as walking, riding a bicycle, or mowing the lawn).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in physical active level | 6 weeks
  Change from physically active levels in METs at 6 weeks

SECONDARY OUTCOMES:
Change in colorectal cancer risk and physical activity coherence | 6 weeks
  Change in understanding of the link between colorectal cancer risk and levels of physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Merced, Merced, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buhi, E. R., Trudnak, T. E., Martinasek, M. P., Oberne, A. B., Fuhrmann, H. J., & McDermott, R. J. (2013). Mobile phone-based behavioural interventions for health: A systematic review. Health Education Journal, 72, 564-583.
- [Background] Cameron LD, Jago L. Emotion regulation interventions: a common-sense model approach. Br J Health Psychol. 2008 May;13(Pt 2):215-21. doi: 10.1348/135910708X288800. Epub 2008 Feb 26. PMID 18302809
- [Background] Durazo, A., & Cameron, L. D. (Manuscript in preparation). A review of cancer risk representations and affect: cancer beliefs and worry as predictors of protection motivation and behavior. Psychological Sciences. University of California, Merced.
- See also: American Cancer Society general information on cancer prevention — http://www.cancer.org